CLINICAL TRIAL: NCT00918008
Title: A 12-Gene Blood-Based Signature for Detecting Metastatic Bladder Cancer
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York Presbyterian Hospital (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-054
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Bladder Cancer
Keywords: URINARY BLADDER; Bladder; Blood sample; Lymph Nodes
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — single blood sample

GROUPS / COHORTS (1):
- Blood sample: the blood sample only collected prior to surgery
  Interventions: Genetic: Blood draw

INTERVENTIONS:
Genetic: Blood draw — The research intervention is the blood sample only collected prior to surgery. Analyses of the data will be made by correlating the gene profile expression with the pathologic finding at surgery and the clinical status of the patients 2 years after surgery.

SUMMARY:
The purposes of this study is to evaluate a new genetic-based test which will identify patients diagnosed with muscle-invasive bladder cancer before their surgery, who might have specific genes, which will increase their chances of recurrence of cancer after their surgery.

Some patients who are diagnosed with bladder cancer and have their had bladder removed, will have a recurrence of cancer sometime after their surgery. This recurrence is usually caused by tumor cells that originated from the bladder tumor and traveled to other parts of the body, which is called metastatic cancer. Some patients are more likely than others to have metastatic disease. This test may help in identifying these patients who might develop metastases from having these specific genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom pelvic lymph node dissection can be performed;
* Any male and/or female, who is ≥18 years of age;
* Pathological diagnosis of urothelial carcinoma of the bladder;
* Localized muscle-invasive disease defined as clinical stage T2-4aN0M0 tumors;
* Did not receive neoadjuvant therapy;
* No radiographic evidence of metastatic disease on CT scans of the abdomen and pelvis, chest x-ray, or bone scan;
* Informed consent before study participation

Exclusion Criteria:

* Prior systemic chemotherapy;
* Prior radiation therapy;
* A history of another ongoing malignancy within the past 5 years other than basal cell carcinoma of the skin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Department of Urology, New York Presbyterian Hospital, Weill Medical College of Cornell University, and from the Department of Surgery, Urology Service at Memorial Sloan-Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Assess the ability of a mononuclear-cell gene signature to predict the presence of metastatic cancer in the regional L.N. of patients with muscle-invasive bladder cancer at the time of cystectomy with PLND for presumed localized muscle-invasive disease. | 2 years

SECONDARY OUTCOMES:
Assess the ability of a mononuclear-cell gene signature, alone or in combination with pathological staging, to predict any metastatic disease w/i 2 yrs of cystectomy with PLND in pts. with clinical organ-confined muscle-invasive bladder cancer staging. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Dalbagni, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm